CLINICAL TRIAL: NCT04911543
Title: An Open-Label Study to Investigate the Regional Brain Kinetics of the Positron Emission Tomography Ligand [18F]-JNJ-70099731 in Healthy Male Participants
Brief Title: A Study to Investigate the Regional Brain Kinetics of the Positron Emission Tomography Ligand [18F]-JNJ-70099731 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: CR108996; 2021-000675-36 (EudraCT Number); 69095897EDI1003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-05-31; First posted 2021-06-03 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A: [18F]-JNJ-70099731 (Experimental): Participants will receive an intravenous (IV) bolus injection of [18F]-JNJ-70099731 on Day 1 of Part A to investigate the total body bio-distribution and measure the radiation dosimetry of [18F]-JNJ-70099731.
  Interventions: Drug: [18F]-JNJ-70099731
- Part B: [18F]-JNJ-70099731 (Experimental): Participants will receive an IV bolus injection of [18F]-JNJ-70099731 on Day 1 of Part B to measure the uptake, distribution, and clearance of [18F]-JNJ-70099731 and to model the tissue specific kinetics of [18F]-JNJ-70099731 in the human brain with the appropriate arterial input function.
  Interventions: Drug: [18F]-JNJ-70099731
- Part C: [18F]-JNJ-70099731 (Experimental): Participants will receive an IV bolus injection of [18F]-JNJ-70099731 on Day 1 of each period of Part C to determine the test-retest variability in the regional brain kinetics and binding properties of [18F]-JNJ-70099731.
  Interventions: Drug: [18F]-JNJ-70099731

INTERVENTIONS:
Drug: [18F]-JNJ-70099731 — [18F]JNJ-70099731 injection will be administered intravenously.

SUMMARY:
The purposes of this study are to measure the whole-body distribution and radiation dosimetry of [18F]-JNJ-70099731 (Part A), to measure the uptake, distribution, and clearance (CL) of [18F]-JNJ-70099731 by Positron Emission Tomography (PET) and to model tissue specific kinetics of [18F]-JNJ-70099731 with the appropriate input function (IF) (Part B), and to measure participant test-retest variability in the distribution of [18F]-JNJ-70099731 by comparing PET scans obtained at least 1 week apart (Part C) in the brain of healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18 and 32 kilogram per meter square (kg/m^2) inclusive
* Participant must be healthy on the basis of physical and neurological examination, medical history, clinical laboratory tests, vital sign (VS), and 12-lead electrocardiogram (ECG) performed at screening. Minor deviations in ECG (example, first-degree atrioventricular block), which are not considered to be of clinical significance to the investigator, are acceptable
* Participant must sign an informed consent form (ICF) indicating that he understands the purpose of and procedures required for the study and is willing to participate in the study
* Part B & Part C only: Participant is willing to allow the investigators to place an arterial catheter in the radial artery. Suitability for arterial catheter placement will be assessed via physical examination (modified Allen Test on both hands). Participant should not be allergic to local anesthetics for catheter placement
* Participant must agree not to donate sperm during the study and for a minimum of 1 spermatogenesis cycle (defined as approximately 90 days) after receiving the last dose of study intervention. If a participant is sexually active with a woman, he should agree to the following: a) If it concerns a woman of childbearing potential and the participant has not had a vasectomy, the participant must agree to use a condom and make sure his female partner is using a highly effective method of birth control during the study and for a minimum of 90 days after the last dose of study intervention; b) If it concerns a woman of nonchild bearing potential or who is pregnant or has been sterilized and the participant has not had a vasectomy, the participant must agree to use a condom for the given period; c) If the participant has had a vasectomy, he should agree to use a condom when being sexually active with a woman of childbearing potential. Contraceptive use by men or women should be consistent with local regulations regarding the use of contraceptive methods for participants participating in clinical studies

Exclusion Criteria:

* Clinically significant abnormal values for hematology, clinical chemistry, coagulation or urinalysis at screening. It is expected that laboratory values will generally be within the normal range for the laboratory, though minor deviations, which are not considered to be of clinical significance to the Principal Investigator, are acceptable
* Clinically significant abnormal physical and neurological examination, VS or 12-lead ECG at screening or before study intervention administration
* History of or current significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, coagulation abnormalities, or other conditions that the Investigator considers should exclude the participant and preclude their ability to participate in study procedures. Participants with a history significant liver or renal disease, or difficulty in urination, which could affect the metabolism and elimination of the radiotracer or radiometabolites should be excluded. Participants with a history of epilepsy or seizures of significance or unexplained black-outs or loss of consciousness should also be excluded
* Exposed to greater than (>)1 millisievert (mSv) of ionizing radiation participating as a participant in research studies and/or at work in the 12 months before the start of this study, to the participant's knowledge
* Serology positive for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibodies or human immunodeficiency virus (HIV) antibodies

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Part A: Normalized Cumulative Activity and Residence Time | Day 1
  Normalized cumulative activity and residence time will be reported.
Part A: Radiation Absorbed Doses for 25 Organs and the Effective Dose (ED) of [18F]-JNJ-70099731 | Day 1
  The tissue radioactivity will be measured per organ for up to 5 hours after injection of [18F]-JNJ-70099731 and corrected for attenuation by computed tomography (CT) transmission scans using positron emission tomography (PET)/CT. These measurements will be used to estimate effective radiation dose per organ and total body.
Part B: Input Function Values kilobecquerel (kBq/cc) for Various Time Points and Tracer Kinetics in Selected Brain Structures | Day 1
  The Distribution of [18F]JNJ-70099731 in brain will be measured by PET/CT scans obtained from the time of injection along with measurement of the tracer input function with arterial samples for intact tracer and metabolites to establish the total and regional compartmental kinetics and volume of distribution.
Part C: Participant Variability in PET Distribution Parameters Over Time | Day 1
  Participant variability in PET distribution parameters over time will be compared between the paired PET scans to assess test-retest variability in the regional brain kinetics and binding properties of [18F]-JNJ-70099731.

SECONDARY OUTCOMES:
Part A, B and C: Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Part A and B: Up to Week 5; Part C: Up to Week 6
  An AE can therefore be any unfavorable and unintended sign (including an abnormal finding), symptom, or disease temporally associated with the use of a medicinal (investigational or non-investigational) product, whether or not related to that medicinal (investigational or non-investigational) product.
Part A, B and C: Number of Participants with Change from Baseline in Treatment Emergent Vital Signs Abnormalities | Part A and B: Baseline, up to Week 5, Part C: Baseline, up to Week 6
  Number of participants with change from baseline in treatment emergent vital signs (Pulse Rate [PR], Systolic Blood Pressure [SBP] and Diastolic Blood Pressure [DBP]) will be assessed.
Part A, B and C: Number of Participants with Change from Baseline in Treatment Emergent Clinical Labs (Chemistry, Hematology, Urinalysis) Abnormalities | Part A and B: Baseline, up to Week 5, Part C: Baseline, up to Week 6
  Number of participants with change from baseline in treatment emergent clinical labs (Chemistry, Hematology, Urinalysis) will be assessed.
Part A, B and C: Number of Participants with Change from Baseline in Treatment Emergent Electrocardiogram (ECG) Abnormalities | Part A and B: Baseline, up to Week 5; Part C: Baseline, up to Week 6
  Number of participants with change from baseline in Heart Rate (HR), Respiratory Rate (RR), QRs Interval, QTc Interval and PR Interval will be measured by ECG.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- UZ Leuven Gasthuisberg, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://www.janssen.com/clinical-trials/transparency